CLINICAL TRIAL: NCT01076153
Title: A Multi-center, Post-Marketing Observational Study to Identify the Recovery Time in Patients With Upper or Lower Respiratory Tract Infections Treated With Klacid MR
Brief Title: Recovery Time in Thai Patients With Upper or Lower Respiratory Tract Infections Treated With Klacid MR
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Savary Om/ Regional Medical Director, Abbott Laboratories
Other Study IDs: P08-331
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Results first posted 2011-06-29 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-06

CONDITIONS: Respiratory Tract Infection
Keywords: Post-marketing observational study; Upper or lower respiratory tract infection; Klacid MR
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Clarithromycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with respiratory tract infection: Thai patients with upper or lower respiratory tract infections on Klacid MR.
  Interventions: Drug: Clarithromycin (Klacid® MR)

INTERVENTIONS:
Drug: Clarithromycin (Klacid® MR) — Klacid MR 500mg (clarithromycin)
  Other Names: Clarithromycin; Klacid MR; Biaxin XL

SUMMARY:
The investigators hypothesize that Klacid modified release (MR) shortens symptom recovery time in Thai patients with upper or lower respiratory tract infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients with upper or lower respiratory tract infection.
* Patient is male or female ≥ 18 years of age.

Exclusion Criteria:

* Known hypersensitivity to or previously intolerant of macrolides.
* Illness severe enough to warrant hospitalization or parenteral therapy.
* Concomitant use of any of the following medications:

  * Drugs metabolized by CYP3A isozyme: alprazolam, astemizole, carbamazepine, cilostazol, cisapride, cyclosporin, disopyramide, ergot alkaloids, lovastatin, methylprednisolone, midazolam, omeprazole, oral anticoagulants (e.g. warfarin), pimozide, quinidine, rifabutin, sildenafil, simvastatin, tacrolimus, terfenadine, triazolam and vinblastine.
  * Drugs metabolized by other isozymes within CYP450 system: phenytoin, theophylline and valproate.
  * Colchicine
  * Digoxin
  * Some antiretrovirals: zidovudine and ritonavir.
* Severe immunodeficiency and chronic disease conditions.
* Renal or hepatic impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients in Thailand
Sampling Method: Non-Probability Sample
Enrollment: 760 (Actual)
Dates: Start 2008-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Savary Om, M.D., Study Director — Abbott
Locations (26):
- Thailand (26):
  - Site Reference ID/Investigator# 27453, Bangkok
  - Site Reference ID/Investigator# 27450, Bangkok
  - Site Reference ID/Investigator# 27448, Bangkok
  - Site Reference ID/Investigator# 22862, Bangkok
  - Site Reference ID/Investigator# 27444, Bangkok
  - Site Reference ID/Investigator# 27445, Bangkok
  - Site Reference ID/Investigator# 27451, Bangkok
  - Site Reference ID/Investigator# 27452, Bangkok
  - Site Reference ID/Investigator# 27449, Bangkok
  - Site Reference ID/Investigator# 27454, Chiang Mai
  - Site Reference ID/Investigator# 27466, Chon Buri
  - Site Reference ID/Investigator# 27465, Chon Buri
  - Site Reference ID/Investigator# 27469, Kanchanaburi
  - Site Reference ID/Investigator# 27455, Nakhon Phanom
  - Site Reference ID/Investigator# 27461, Nakhon Ratchasima
  - Site Reference ID/Investigator# 27462, Nakhon Ratchasima
  - Site Reference ID/Investigator# 27463, Nakhon Ratchasima
  - Site Reference ID/Investigator# 27457, Nong Khai
  - Site Reference ID/Investigator# 27458, Nong Khai
  - Site Reference ID/Investigator# 27467, Rayong
  - Site Reference ID/Investigator# 27470, Songkhla
  - Site Reference ID/Investigator# 27472, Surat Thani
  - Site Reference ID/Investigator# 27471, Surat Thani
  - Site Reference ID/Investigator# 27459, Ubonratchathani
  - Site Reference ID/Investigator# 27456, Udon Thani
  - Site Reference ID/Investigator# 27464, Uttaradit

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 760 participants were enrolled in the study. 694 were analyzed as 66 participants had protocol deviations (some more than 1): Age less than 18 years (22), took excluded drugs (17), took Klacid more than 14 days (16), took Klacid less than 5 days (11), added 250 mg Klacid to Klacid MR (5), and used injectable drugs (3).
Groups:
- Klacid MR: Male or female Thai adults with upper and/or lower respiratory tract infections taking Klacid (clarithromycin) modified release (MR) 500 mg according to the Prescribing Information.
Period: Overall Study
Arm/Group | Klacid MR
Started | 760
Completed | 749
Not Completed | 11
Not completed — Symptoms improved/resolved | 10
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Klacid MR: The per-protocol population (694 participants) of male or female Thai adults with upper and/or lower respiratory tract infections on Klacid MR.
Arm/Group | Klacid MR
Number analyzed (Participants) | 694
Age Continuous [Mean (Standard Deviation); unit: years] — Based on per-protocol population (694 participants).
  years | 41.16 (14.22)
Age, Customized [Number; unit: participants] — Based on per-protocol population (694 participants).
  participants
    18 to 20 years | 28
    21 to 30 years | 154
    31 to 40 years | 204
    41 to 50 years | 141
    51 to 60 years | 102
    Over 60 years | 65
Sex: Female, Male [Count of Participants; unit: Participants] — Based on per-protocol population (694 participants).
  Participants
    Female | 404
    Male | 290
Region of Enrollment [Number; unit: participants] — Based on per-protocol population (694 participants).
  participants
    Thailand | 694
Diagnosis [Number; unit: participants] — Participant diagnosis at study entry for the per-protocol population (694 participants).
  participants
    Upper respiratory tract infection | 510
    Lower respiratory tract infection | 165
    Both upper and lower respiratory tract infections | 19
Risk factor: Smoking status [Number; unit: participants] — Whether or not participants smoked cigarettes for the per-protocol population (694 participants).
  participants
    Participant was a smoker | 164
    Participant did not smoke | 530

OUTCOME MEASURES:

1. Primary Outcome: Average Time From Baseline to Recovery From Cough and Other Symptoms
Description: Study participants were seen at an initial visit (baseline) and received Klacid treatment for 5 to 14 days. A medical appointment (visit or phone call) was made 6 to 14 days after the first visit. Participants' symptoms were rated using one of the following categories: resolved, improved, not changed, or worse. Associated dates were also recorded. Symptoms included, but were not limited to, cough, fever, and sore throat. Recovery was defined as the disappearance of all signs and symptoms of infection.
Time Frame: Baseline to 14 days
Population: The per-protocol population consisted of 694 participants as 66 participants were excluded for protocol deviations (some more than 1): Age less than 18 years (22), took excluded drugs (17), took Klacid more than 14 days (16), took Klacid less than 5 days (11), added 250 mg Klacid to Klacid MR (5), and used injectable drugs (3).
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Klacid MR (Total Number Recovered): Male or female Thai adults with upper and/or lower respiratory tract infections on Klacid MR who were in the recovered population.
- Klacid MR (URTI, Recovered): Participants in the recovered population who had a diagnosis of upper respiratory tract infection (URTI) at study entry.
- Klacid MR (LRTI, Recovered): Participants in the recovered population who had a diagnosis of lower respiratory tract infection (LRTI) at study entry.
- Klacid MR (URTI and LRTI, Recovered): Participants in the recovered population who had a diagnosis of both upper and lower respiratory tract infections at study entry.
Arm/Group | Klacid MR (Total Number Recovered) | Klacid MR (URTI, Recovered) | Klacid MR (LRTI, Recovered) | Klacid MR (URTI and LRTI, Recovered)
Number analyzed (Participants) | 658 | 491 | 148 | 19
Days | 7.06 (2.65) | 6.76 (2.11) | 7.82 (3.75) | 9.05 (3.08)

2. Secondary Outcome: Number and Type of Adverse Events
Description: Adverse events were collected during the course of the study up to 30 days or 5 half-lives following the last dose of Klacid. The number of participants experiencing a serious or non-serious adverse event is summarized. See the Reported Adverse Event section for details.
Time Frame: Baseline to 14 days
Population: The safety population included all participants who took at least 1 dose of Klacid.
Measure: Number; unit: Events
Arm/Group | Klacid MR
Number analyzed (Participants) | 760
Events
  Serious Adverse Events | 0
  Non-serious Adverse Events | 7

ADVERSE EVENTS:
Time Frame: All adverse events that occurred during the course of the study were reported in detail on case report forms. Adverse events occurring during the study were reported up to 30 days or 5 half-lives after the last dose of Klacid MR.
Arm/Group | Klacid MR
Serious Adverse Events (participants affected / at risk) | 0/760
Other Adverse Events (participants affected / at risk) | 5/760
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Klacid MR (N=760)
Dysgeusia (Gastrointestinal disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Muscle strain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.